CLINICAL TRIAL: NCT00189397
Title: Azathioprine Versus Corticosteroids for the Treatment of Parthenium Dermatitis
Brief Title: Azathioprine Versus Corticosteroids in Parthenium Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD 358; I 358
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Parthenium Dermatitis
Keywords: Parthenium dermatitis
MeSH Terms: conditions — Parthenium dermatitis | interventions — Azathioprine; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: azathioprine and corticosteroids for Parthenium dermatitis

SUMMARY:
The dermatitis caused by the substances which come in contact with the skin is known as contact dermatitis. When such a reaction is caused by the agents suspended in the air, it is called air-borne contact dermatitis (ABCD). Parthenium hysterophorus at present is the commonest cause of ABCD in India though in some cases other plants have also been found to cause ABCD. Parthenium dermatitis is one of the major health problems in dermatology in our country. Though it has very little mortality, the disease normally continues to persist with variable remissions and relapses causing great distress and morbidity. Corticosteroids, topical and systemic have been the mainstay of the treatment so far. Therefore, the patients with ABCD who have to take corticosteroids for long periods of time tend to develop severe and sometimes irreversible side effects of the therapy. Azathioprine is an immunosuppressive drug which acts by inhibiting the T lymphocytes. In our previous studies we have been able to induce remissions in these patients with azathioprine used as daily as well as monthly bolus dose, without having to use systemic corticosteroids. The side effect with azathioprine in these studies were almost absent.

We have therefore planned to study the therapeutic efficacy of azathioprine weekly pulse doses versus daily azathioprine in achieving remissions in patients having Parthenium dermatitis and to monitor the side effects of both the regimens.

DETAILED DESCRIPTION:
Detailed research plan Clinical evaluation About 60 clinically diagnosed adult patients having Parthenium dermatitis will be taken up for the study. Pregnant females and lactating mothers will be excluded. All the patients will be patch tested with the standardised aqueous extract of Parthenium hysterophorus to confirm the diagnosis and those showing positive patch test reactions to standardised extract will be tested further with serial dilutions of the antigens to determine the titre of contact hypersensitivity (TCH).20 Antibodies do not have any role in this disease therefore the estimation of immunoglobulins will not be done. The diagnosis will be done by patch test. It will be a randomised, clinically study where the patients will be randomly treated with azathioprine 300 mg per week or azathioprine 100 mg a day orally along with topical clobetasol propionate 0.05% w/w and oral cetirizine hydrochloride 10 mg daily for symptomatic relief. No other drugs including the medicines of alternate system will be given for the dermatitis. Clinical evaluation of the patients will be undertaken every four weeks. This will be continued for six months. After 6 months the treatment will be stopped and the patients will be followed up for another 6 months. The graphic record of the disease activity and the treatment will be maintained. In addition, each patient will be evaluated for the side effects of these regimens clinically as well as by the laboratory parameters as per the proforma enclosed, especially haemoglobin, total blood count, differential count, platelets, serum bilirubin, serum alkaline phosphate, serum transaminases, serum electrolytes, serum creatinine, blood urea, blood sugar, urine routine and microscopy and stool examination for occult blood. These tests will be carried out before starting the therapy and then repeated every month during the follow up period. Chest X-ray electrocardiogram and TCH will also be done before the therapy and then at six months unless otherwise required. At the end of the study period, a final evaluation based on the change in severity of the dermatitis, changes in the titre of contact hypersensitivity and the side effects of the drugs will be made. Statistical analysis using chi-square test will be done.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients having ABCD, as shown by the clinical manifestations and positive patch tests with Parthenium, who are willing to participate in the study.

Exclusion Criteria:

* Patients below the age of 18 years
* Pregnant and lactating women.
* Patients whose baseline investigations reveal hematological abnormalities or abnormalities of liver or renal function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2005-10 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Clinical remission and side effects

SECONDARY OUTCOMES:
Duration of remission

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal K Verma, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Department of Dermatology, AIIMS, New Delhi, National Capital Territory of Delhi, India